CLINICAL TRIAL: NCT07220317
Title: A Clinical Evaluation of Orthodontic Tooth Movements in Mixed Dentition
Brief Title: This Study Will Examine Shortened Treatment Wear Time for Patients With Mixed Dentition Using AirFlex Aligner, Sequential Dental Aligners.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoFX (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-370
Record Dates: First submitted 2025-10-09; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Mixed Dentition Using Sequential Dental Aligners
Keywords: mixed dentition; dental aligners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental: Short wear (Experimental): Short wear
  Interventions: Device: Sequential Aligners

INTERVENTIONS:
Device: Sequential Aligners — Treatment with sequential aligners in a shortened wear time with mixed dentition.

SUMMARY:
This study will examine shortened treatment wear time for patients with mixed dentition using sequential dental aligners. Using the existing AirFlex aligner design that patients with permanent dentition use, it may be possible to reduce the wear time and still provide dental realignment in an adequate treatment period for patients with mixed dentition. The Airflex aligner will be tested for a 9-12-hour patient wear time.

DETAILED DESCRIPTION:
The primary intervention is the change in active wear time. In current practice, sequential aligners are prescribed to be worn approximately 20 to 22 hours per day. In this study, the prescribed wear time will be reduced to 9 - 12 hours per day.

This study is intended to demonstrate effectiveness of AirFlex aligners, which have a reduced wear time compared to traditional aligners, in mixed dentition subjects. The study will be conducted using AirFlex aligners, which are currently cleared for treatment of patients with permanent dentition.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 7 to 21 years old
* Mixed dentition, as defined by the presence of at least one primary tooth present at the start of orthodontic treatment
* No untreated cavities
* Good Periodontal composition as determined by dental exam

Exclusion Criteria:

* Skeletal discrepancies requiring surgery
* Is currently undergoing dental/orthodontic work
* Has dental prosthesis/implants that will interfere with projected tooth movement
* Ongoing use of medication affecting tooth movement or bone formation (NSAIDS, Steroids, Bisphosphonates, Levothyroxine, Teriparatides, etc.)
* Is currently pregnant or plans to become pregnant during treatment
* Current smoker or tobacco use within 2 years
* Presence of systemic diseases that could interfere with treatment
* Moderate or significant periodontal disease
* Any other physical exam finding that precludes participation

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will assess the tooth movements (torque, extrusion, rotation, translation, intrusions, and tipping), ensuring that final dentition is within 0.3 mm of the intended position. | 16 weeks

IPD SHARING:
Plan to Share IPD: Undecided